CLINICAL TRIAL: NCT02928497
Title: Assessment of the WATCHMAN™ Device in Patients Unsuitable for Oral Anticoagulation (ASAP-TOO)
Brief Title: Assessment of the WATCHMAN™ Device in Patients Unsuitable for Oral Anticoagulation
Acronym: ASAP-TOO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S2317
Record Dates: First submitted 2016-10-05; First posted 2016-10-10 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: Non-valvular atrial fibrillation; Left atrial appendage
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- WATCHMAN (Device) (Experimental): WATCHMAN LAAC Device implant including modified post-implant drug regimen.
  Interventions: Device: WATCHMAN LAAC Device Implant
- Control (Active Comparator): Single antiplatelet therapy or no therapy (Control) at the discretion of the study physician for the duration of the trial.
  Interventions: Drug: Single Antiplatelet Therapy or No Therapy (Control)

INTERVENTIONS:
Device: WATCHMAN LAAC Device Implant — WATCHMAN LAAC Implant
  Arms: WATCHMAN (Device)
Drug: Single Antiplatelet Therapy or No Therapy (Control) — Single Antiplatelet Therapy or No Therapy at the discretion of the study physician.
  Arms: Control

SUMMARY:
The purpose of this study is to establish the safety and effectiveness of the WATCHMAN™ Left Atrial Appendage Closure (LAAC) Device, including the post-implant medication regimen, for subjects with non-valvular atrial fibrillation who are deemed not to be eligible for anti-coagulation therapy to reduce the risk of stroke.

DETAILED DESCRIPTION:
The ASAP-TOO study is a prospective, randomized, multi-center, global investigation to establish the safety and effectiveness of the WATCHMAN Device for subjects with non-valvular atrial fibrillation who are deemed not suitable for anti-coagulation therapy to reduce the risk of stroke.

Subjects will be randomized in a ratio of 2 Device to 1 Control to receive the WATCHMAN LAA closure device (Device) or the control treatment of single antiplatelet medication or no medication at the discretion of the study physician (Control). All randomized subjects will follow the protocol required tests and assessments at each scheduled follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* The subject is of legal age to participate in the study per the laws of their respective geography.
* The subject has documented paroxysmal, persistent, permanent or long-term/longstanding persistent non-valvular atrial fibrillation (i.e., the subject has not been diagnosed with rheumatic mitral valvular heart disease).
* The subject has a calculated CHA2DS2-VASc score of 2 or greater.
* The subject is deemed by two study physicians to be unsuitable for oral anticoagulation.
* The subject is deemed by a study physician to be suitable for the defined protocol pharmacologic regimen of aspirin and clopidogrel therapy following WATCHMAN Closure Device implant.
* The subject or legal representative is able to understand and willing to provide written informed consent to participate in the trial.
* The subject is able and willing to return for required follow-up visits and examinations.

Exclusion Criteria:

* The subject is unable or unwilling to return for required follow-up visits and examinations.
* The subject had or is planning to have any invasive cardiac procedure within 30 days prior to randomization (e.g., cardioversion, ablation).
* The subject is planning to have any cardiac or non-cardiac invasive or surgical procedure that would necessitate stopping or modifying the protocol required medication regimen within 90 days after the WATCHMAN Closure Device implant (e.g., cardioversion, ablation, cataract surgery).
* The subject had a prior stroke (of any cause) or TIA within the 30 days prior to randomization.
* The subject had a prior BARC type 3 or 4 bleeding event within the 14 days prior to randomization. Lack of resolution of related clinical sequelae, or planned and pending interventions to resolve bleeding/bleeding source, are a further exclusion regardless of timing of the bleeding event.
* The subject has a history of atrial septal repair or has an ASD/PFO device.
* The subject has an implanted mechanical valve prosthesis in any position.
* The subject suffers from New York Heart Association Class IV Congestive Heart Failure.
* The subject has LVEF < 30%.
* The subject is of childbearing potential and is, or plans to become pregnant during the time of the study (method of assessment upon study physician's discretion).
* The subject is currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance should be brought to the attention of the sponsor to determine eligibility.
* The subject has a life expectancy of less than two years.
* The subject has a known or suspected hypercoagulable state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Primary 7-Day Device/Procedural Safety Endpoint | 7 days
  The primary safety endpoint is the 7-day combined rate of death, ischemic stroke, systemic embolism and complications requiring major cardiovascular or endovascular intervention.
Primary Efficacy Endpoint - time to first event of ischemic stroke or systemic embolism. | 5 years
  The primary efficacy endpoint is the comparison of time to first event of ischemic stroke and systemic embolism.

SECONDARY OUTCOMES:
Secondary Endpoint - Composite of All Stroke and Cardiovascular or Unknown Death | 5 years
  The occurrence of stroke (including ischemic and/or hemorrhagic), cardiovascular death (cardiovascular and/or unexplained cause) and systemic embolism
Secondary Endpoint - Major Bleeding | 5 years
  The occurrence of major bleeding (defined as a BARC Type 3 or 5 event)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Saw, MD, Principal Investigator — Vancouver General Hospital; Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Maurice Buchbinder, MD, Principal Investigator — Stanford University
Locations (92):
- United States (71):
  - Grandview Medical Center, Birmingham, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Scripps Memorial Hospital, La Jolla, California
  - Cedars - Sinai Medical Center, Los Angeles, California
  - Sharpe Chula Vista Medical Center, San Diego, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - St. John's Health Center, Santa Monica, California
  - North Colorado Medical Center, Greeley, Colorado
  - St. Anthony Hospital, Lakewood, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Delray Medical Center, Delray Beach, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Bay Area Cardiology Associates, Tampa, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Edward Hospital, Naperville, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St. John's Hospital, Springfield, Illinois
  - St. Vincent's Hospital, Indianapolis, Indiana
  - Heart Group at Deaconness Hospital, Newburgh, Indiana
  - Mercy Hospital Medical Center, West Des Moines, Iowa
  - Kansas City Cardiac Arrhythmia Research, Overland Park, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Maine Medical Center, Portland, Maine
  - Union Memorial Hospital, Baltimore, Maryland
  - Southcoast Physicians Group, Fall River, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Foundation, Rochester, Minnesota
  - Centracare Heart and Vascular, Saint Cloud, Minnesota
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Mercy Research, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - The Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Catholic Medical Center, Manchester, New Hampshire
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - St. Barnabas Medical Center, Newark, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Northwell Health, Staten Island, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Summa Health System, Akron, Ohio
  - Aultman Hospital, Canton, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - OhioHealth Research and Innovation Institute - Riverside Methodist Hospital, Columbus, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - UPMC Heart and Vascular Institute Harrisburg, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Saint Thomas Health, Nashville, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - University of Texas Houston Health Science Center, The Woodlands, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - CHI Franciscan Health System, Tacoma, Washington
  - PeaceHealth Southwest Medical, Vancouver, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
  - Aspirus Heart and Vascular Institute - Research and Education, Wausau, Wisconsin
- Belgium (2):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - ZNA Middelheim, Antwerp
- Canada (3):
  - Ottawa Heart Institute, Ottawa
  - Institut universitaire de Cardiologie et de Pneumologie de Quebec, Ste-foy
  - Vancouver General Hospital, Vancouver
- Na Homolce Hospital, Prague, Czechia
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet Copenhagen, Copenhagen
- Germany (5):
  - Universitaetsklinikum Dusseldorf, Düsseldorf
  - St.Johann Nepomuk Katholisches Hospitalvereinigung Thüringen GmbH, Erfurt
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Cardiologicum Hamburg Praxis Wandsbek, Hamburg
  - Herzzentrum Universität Leipzig, Leipzig
- Fondazione Toscana Gabriele Monasterio, Massa, Italy
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede
  - St. Antonius Ziekenhuis, Nieuwegein
- United Kingdom (5):
  - Royal Victoria Hospital, Belfast
  - Royal Sussex County Hospital, Brighton
  - Guys and St. Thomas NHS Foundation Trust, London
  - The Brompton Hospital, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alomar M, Fradley MG. Electrophysiology Translational Considerations in Cardio-Oncology: QT and Beyond. J Cardiovasc Transl Res. 2020 Jun;13(3):390-401. doi: 10.1007/s12265-019-09924-y. Epub 2019 Oct 31. PMID 31673900